CLINICAL TRIAL: NCT06585657
Title: Clinical Study on Brain Visual Perception Training for Prevention and Control of Myopia in Children with Premyopia
Brief Title: Brain Visual Perception Training for Prevention and Control of Premyopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: QX-2024-A-011
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Visual Function; Myopia Progressing
Keywords: brain visual perception training; premyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- brain visual perception training group (Experimental): Conduct brain visual perception training through a visual training system to improve binocular visual balance. Train 2 projects per day, each lasting 10 minutes.
  Interventions: Device: brain visual perception training group
- control group (No Intervention): no intervention

INTERVENTIONS:
Device: brain visual perception training group — Conduct brain visual perception training through a visual training system to improve binocular visual balance. Train 2 projects per day, each lasting 10 minutes.
  Arms: brain visual perception training group

SUMMARY:
The goal of this clinical trial is to investigate whether brain visual perception training can effectively prevent myopia in children with pre myopia. It will also learn about the safety of brain visual perception training.

The main questions it aims to answer are: Does brain visual perception training slow down the growth of axial length? What medical issues may participants encounter when using the brain visual perception training system? Researchers will compare participants who receive brain visual perception training with a control group to see if the training group can delay the onset of pre myopia in children Participants will: The training group will receive 20 minutes of brain visual perception training once a day for a period of one year. Follow up check ups at the hospital every 3 months. Keep a diary of the values of axial length and refractive diopter.

ELIGIBILITY:
Inclusion Criteria:

Children aged 6-10 years with premyopia, defined as a cycloplegic spherical equivalent refraction (SER) of the more myopic eye in the range of -0.50 to 0.75 (inclusive) diopters (D) and having at least 1parent with an SER in either eye of -3.00D or less.

Exclusion Criteria:

Children have astigmatism of 1.50D or more, anisometropia of 1.50 D or more, strabismus and other ocular abnormalities, any systemic diseases, or a history of any myopia interventions.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 156 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
changes in axial length after 1 year | 1 year after the baseline
  the difference in the changes of axial length between the intervention group and the control group

SECONDARY OUTCOMES:
changes in cycloplegic spherical equivalent after 1year | 1 year after the baseline
  the difference in the changes of cyclopegic spherical equivalent between the intervention group and the control group

IPD SHARING:
Plan to Share IPD: No